CLINICAL TRIAL: NCT01743144
Title: Study the Possible Effects of Intraoperative Intravenous Magnesium Sulphate Infusion on the Incidence of Sevoflurane Induced Emergence Agitation in Children Undergoing Adenotonsillectomy
Brief Title: Magnesium Sulphate and Sevoflurane Induced Emergence Agitation in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Collaborators: anesthesia department (Ambiguous); faculty of medicine (Ambiguous)
Responsible Party: Principal Investigator, Abeer Ahmed, lecturer of anesthesia, faculty of medicine, cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: N-40-2012
Record Dates: First submitted 2012-11-18; First posted 2012-12-06 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Emergence Delirium; Postopertive Delirium; Emergence Agitation in Children
Keywords: emergence agitation in children; sevoflurane; general anesthesia; magnesium sulphate
MeSH Terms: conditions — Emergence Delirium | interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Magnesium sulphate (Active Comparator): Magnesium sulphate (MgSO4) 10% solution is going to be used, an initial MgSO4 bolus dose 30mg/kg (i.e. 0.3mL/kg) will be infused over 10 minutes after endotracheal intubation. This will be followed by a continuous infusion of 10 mg/kg/hr (i.e. 0.1 ml/kg/h). Infusion will continue during the entire intraoperative course and will be terminated with the discontinuation of sevoflurane
  Interventions: Drug: Magnesium Sulfate
- normal saline (Placebo Comparator): normal saline (NaCl 9%) is going to be used, an initial normal saline bolus dose 0.3ml/kg will be infused over 10 minutes after endotracheal intubation. This will be followed by a continuous normal saline infusion of 0.1 ml/kg/h. Infusion will continue during the entire intraoperative course and will be terminated with the discontinuation of sevoflurane
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Magnesium Sulfate — Magnesium sulphate (MgSO4) 10% solution is going to be used, an initial MgSO4 bolus dose 30mg/kg (i.e. 0.3mL/kg) will be infused over 10 minutes after endotracheal intubation. This will be followed by a continuous infusion of 10 mg/kg/hr (i.e. 0.1 ml/kg/h). Infusion will continue during the entire intraoperative course and will be terminated with the discontinuation of sevoflurane
  Arms: Magnesium sulphate
Drug: normal saline — normal saline (NaCl 9%) is going to be used, an initial normal saline bolus dose 0.3ml/kg will be infused over 10 minutes after endotracheal intubation. This will be followed by a continuous normal saline infusion of 0.1 ml/kg/h. Infusion will continue during the entire intraoperative course and will be terminated with the discontinuation of sevoflurane
  Arms: normal saline

SUMMARY:
Rationale:

Pediatric Adenotonsillectomy is a common procedure of brief performed on a day-case basis, in which rapid recovery with safe airway after extubation is crucial. Sevoflurane is considered the inhaled anesthetic of choice in such procedures, however it has been reported that emergence agitation (EA) is a frequent complication in 30-80% of children receiving sevoflurane general anesthesia. The possible effect of magnesium sulphate on decreasing the incidence of EA in children was not adequately investigated.

Objective:

To assess the possible effects of intraoperative intravenous magnesium sulphate (MgSO4) infusion on the incidence of sevoflurane-induced EA in children undergoing adenotonsillectomy.

Study population and sample size:

Children 4-7 years, ASA physical status I or II, undergoing Adenotonsillectomy under sevoflurane general anesthesia. 64 patients (32/group) is required to detect a significance difference of 40% in the incidence of agitation between two groups, with a power of 80% and alpha error of 5%.

Study design:

A double blind, randomized, placebo controlled study.

Method:

In the placebo group, a normal saline bolus dose 0.3ml/kg will be iv infused followed by a continuous infusion of 0.1 ml/kg/h. In the MgSO4 group, a MgSO4 bolus dose 0.3mL/kg will be iv infused followed by a continuous infusion of 0.1 ml/kg/h. infusion terminated by the end of surgery. Post operative emergence agitation will be assessed by using the Pediatric Anesthesia Emergence Delirium scale.

Possible risks:

Drug side effects such as facial warmth, flushing, dry mouth, and malaise.

Outcome parameters:

The primary outcome: incidence of sevoflurane-induced EA measured using the Pediatric Anesthesia Emergence Delirium (PEAD). Secondary outcome: postoperative pain and rescue analgesic requirements, perioperative hemodynamics, durations of recovery, postoperative complications

Statistical analysis plan:

Student's t-test or Mann Whitney-U and Chi square or Fisher's exact tests will be used as appropriate. The possible relationship between EA and pain scores will be evaluated with the use of Spearman's rank correlation coefficient

Time plan:

6-9 months.

ELIGIBILITY:
Inclusion Criteria:

Children 4-7 years, ASA physical status I or II, undergoing Adenotonsillectomy will be included in the study.

Exclusion Criteria:

* The study will exclude children with behavioral changes, physical developmental delay and children on treatment with sedative or anticonvulsant. Also children with pre-existing renal disease or cardiovascular diseases will be excluded.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
change from baseline of sevoflurane induced emergence agitation(EA) at 2 hours postoperative by using Pediatric Anesthesia Emergence Delirium (PEAD) score | on arrival to post anesthesia care unit (PACU) as baseline , then every 10 minutes up to 2 hours postoperatively

SECONDARY OUTCOMES:
postoperative pain which is going to be assessed by the well established behavior pain scale "Children's Hospital Eastern Ontario Scale" (CHEOPS) | on arrival to post anesthesia care unit (PACU) as baseline , then every 10 minutes up to 2 hours postoperatively

OTHER OUTCOMES:
post operative rescue analgesic requirements, perioperative hemodynamic variables, durations of recovery, hospital stay and postoperative complications (vomiting, laryngospasm, bronchospasm, or bleeding from surgical site). | for 2 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdulatif, Anesthesia Professor, Study Chair — Anesthesia department-Faculty of medicine-Cairo University
Locations (1):
- Anesthesia department - Faculty of medicine- Cairo University, Cairo, Cairo Governorate, Egypt